CLINICAL TRIAL: NCT02368392
Title: National Cardiac Arrest Survey of Sri Lanka
Brief Title: National Cardiac Arrest Survey
Acronym: NCAS
Status: Completed | Type: Observational
Sponsor: Ministry of Health, Sri Lanka (Other Government)
Collaborators: National Intensive Care Surveillance (Other); Mahidol Oxford Tropical Medicine Research Unit (Other); Government Medical Officers Association of Sri Lanka (Unknown)
Responsible Party: Principal Investigator, Pubudu De Silva, Consultant Community Physician, Ministry of Health, Sri Lanka
Other Study IDs: NCAS
Record Dates: First submitted 2015-02-14; First posted 2015-02-23 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: In-hospital Cardiac Arrest
Keywords: in-hospital cardiac arrest; quality of life after cardiac arrest; survival after cardiac arrest; resources for cardiac arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cardiac Arrest: Those who get in-hospital cardiac arrests
  Interventions: Other: Exposure for cardiac arrests
- Non Cardiac Arrest: Those who do not get in-hospital cardiac arrest
  Interventions: Other: Exposure for cardiac arrests

INTERVENTIONS:
Other: Exposure for cardiac arrests — There is no particular intervention. This study merely observes the occurrence of cardiac arrests

SUMMARY:
The aim of this study is to describe incidence of "in-hospital" deaths and outcomes after attempted cardiac arrest resuscitation, availability of resuscitation equipment and medical staff training in state Hospitals of Sri Lanka.

DETAILED DESCRIPTION:
4 General objective To describe incidence of "in-hospital" deaths, outcomes after attempted cardiac arrest resuscitation and availability of resuscitation equipment in Sri Lankan state Hospitals.

4.1 Specific objectives

* To describe the incidence of in-hospital deaths in state sector Hospitals in Sri Lanka.
* To describe the availability of resources for cardiac arrest management in these settings.
* To describe the incidence of attempted resuscitation after cardiac arrests.
* To describe the immediate outcomes after attempted resuscitation for cardiac arrests.
* To describe the ICU, Hospital and 30 day post discharge outcomes of these patients
* To describe the health related quality of patients who survived to 1 year

  5 Methodology 5.1 Study one 5.1.1 Study design One week cross-sectional study

5.1.2 Study setting In all state sector Hospitals with (Base Hospitals and above)

5.1.3 Administrative process Once ethical review process has been completed, The Hospital Directors/Medical Superintendent (and through them the Hospital Consultants) will be officially informed of the study by the office of the Deputy Director General (Education, Training and Research) (DDG ET&R) at the Ministry of Health.

Medical Officers will be nominated for the study through the same office. A small financial incentive will be provided for these Doctors during this study period (as below). The investigators will also seek permission from the Steering committee of National Intensive Care Surveillance to obtain ICU admission, outcome and follow-up data for IHCA patients from the NICS database.

5.1.4 Study population All patients who died in-hospital or those on whom CPR was attempted within the time period of the study.

5.1.4.1 Exclusions criteria

* Dead on arrival at Hospital
* Neonate (less than 28 days)

5.1.5 Study sample Entire population

5.1.6 Study period One week period in July/August 2014

5.1.7 Sample size One week period will be studied

5.1.8 Sampling method Not applicable

5.1.9 Data collection tools During the study period, nominated and pre-trained medical officers from each Hospital will complete a questionnaire using an online form on a daily basis. The data collector will interview each Ward Sister, House Officer or senior nurse twice (around 7 am and 7 pm) daily. Non- ward areas such as operating theatres, emergency rooms will also be covered. This process will be piloted in five hospitals prior to the study to fine tune the process.

5.1.9.1 Data validation Death register in the ward/mortuary or in the Matron's office will be used to validate the data collected on Hospital deaths and any discrepancies resolved. Random validation of the data collected at Hospital level will be done centrally on a daily basis during the one-week period.

ICU admission reasons will also be collected from all ICUs during this period to detect ICU admissions due to in-hospital cardiac arrests, which can also be used as a method of validation.

5.1.10 Study variables The following will be collected daily during the one week period

* Number of in-ward deaths
* Number of attempted resuscitations
* Number of successful resuscitations and their subsequent locations
* Number admitted to ICU (name and BHT number) following resuscitation and location of the ICUs
* Total number of in-ward patients at midnight, daily, during the study period.
* In addition at the beginning of the study period the facilities available for resuscitation will be collected at ward/theatre against a standard resuscitation council equipment checklist. The staff participation in previous resuscitation training will be gathered anonymously at the same time. This information will only be collected once.

5.2 Study two 5.2.1 Study design Longitudinal study

5.2.2 Study setting All Intensive Care Units to which the patients successfully resuscitated have been admitted.

5.2.3 Study period From the beginning of the study period of study 1 above, and until 30 days after ICU discharge for the last patient admitted to an ICU after successful resuscitation, up to a maximum of 90 days from the start of the study period.

5.2.4 Sample size All patients admitted to an ICU after successful resuscitation from study 1 above, will be included. We are unable to estimate a sample size for this study as the number of patients admitted after cardiac arrests over this period is not known. The purpose of this part of the study is to actually know what number of patients are admitted to ICU after resuscitation and what their outcomes are. No causative association is proposed as an product of this part of the study.We have selected a one-week recruitment period as this is a national study and we feel this is a feasible duration for us.

5.2.5 Sampling method All patients who had successful resuscitation and were admitted to ICU in study 1, will be included.

5.2.6 Data collection tools The data will be gathered, after appropriate permission has been sought, as above, from the National Intensive Care Surveillance (NICS) database. No new data will need to be gathered from these ICUs. If the ICU is not part of the NICS network, we will follow up these resuscitated patients in these non-NICS ICUs. Health related Quality of Life,neurological and disability status of these patients will be reviewed using SF-12, EQ-5Dand MRS from those who survived to 1 year.

5.2.7 Study variables The following data will be collected for each eligible patient using the National Intensive Care Surveillance database where the ICU is part of the network.

* Outcomes at ICU discharge
* Outcomes at Hospital discharge
* Outcomes at 30 day post discharge In the non-NICS ICUs we will determine ICU outcomes by contacting the ICUs at least once a week. We will also determine hospital and 30 days outcome by obtaining a contact telephone number of the patient or the next of kin. This is similar to the methodology we currently employ for patients admitted to NICS ICUs.
* Health related Quality of Life, neurological and disability status of patients who survived at 6 months and up to 1 year

  6 Statistical analysis: Data will be analyzed using Statistical Package for Social Sciences 18 and Stata 13.

Discrete variables are expressed as counts (percentage) and continuous variables as means (± standard deviations (SD) and median (inter quartile range (IQR)). For description of variables standard descriptive statistics will be used. For comparison of continuous variables t test will be used while chi square will be used to compare discrete variables.

Multivariate logistic regression analysis will be used to describe the prevalence of selected factors as antecedents or contributory features of cardiac arrests.

7 Ethics 7.1 Consent: Permission will be taken from the relevant Authorities of the Ministry of Health and Hospitals as described in detail above. Personal identifier data of patients will not be collected except for Name, BHT number, address and telephone number of those successfully resuscitated. The investigators and data collectors will not come in direct contact with the patients except when determining 30 day outcome.

7.2 Risks to the patient: There are no obvious risks to patient.

7.3 Benefits: Potential benefits are many at individual patient level, Hospital level and national level. The study will enable quantification of the burden of recognized cardiac arrests, their outcomes and possible antecedent/contributory factors to enable the formulation of concrete strategies to improve care.

7.4 Confidentiality: Data extraction sheet will be completed only by the nominated medical officers or by the proposed expert committee. Data will be stored in a computer and only the authorized personal will have access to this information and the information will be password protected and backed up.

7.5 Dissemination of information: The findings will be disseminated in the form of abstracts submitted for scientific session, journal articles and presentations. They may be used for local or national guideline preparation.

7.6 Beneficiaries: There are three main categories of beneficiaries. The Ministry of Health benefits from information by knowing the ground situation and being able to plan and direct the donors where improvement are needed both in resources as well as capacity building. The staff benefits by being able to identify areas of improvement in the services given for IHCA and resuscitation and thus has the opportunity to improve the skills on resuscitation. Thus data can be used to develop services and the human resources in improving IHCA management and patient out come.

ELIGIBILITY:
Inclusion Criteria:

* All admissions to state hospitals in Sri Lanka

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitting to state hospitals in Sri Lanka
Sampling Method: Probability Sample
Enrollment: 537 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 day
  Mortality 30 days after cardiac arrest

SECONDARY OUTCOMES:
ICU admission | 30 day
  ICU admissions following cardiac arrests
Quality of Life | 1 year
  Quality of life of survivors of cardiac arrests
Survival | 1 year
  1 year survival after cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Rashan Haniffa, MBBS, FRCA, Study Chair — Mahidol Oxford Tropical Medicine Research Unit; Saroj Jayasinghe, MD, FRCP, Study Chair — University of Colombo
Locations (1):
- National Intensive Care Surveillance, Colombo, Sri Lanka